CLINICAL TRIAL: NCT05136040
Title: Comparison Of The Effects Of Two Different Low-Doses Of Isobaric Bupivacaine On Intraoperative Hemodynamics In Spinal Anesthesia During Cesarean Section: A Randomized Controlled Trial
Brief Title: Low-Doses Of Isobaric Bupivacaine On Intraoperative Hemodynamics In Spinal Anesthesia During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B.30.2.ATA.0.01.00
Record Dates: First submitted 2021-10-21; First posted 2021-11-26 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Cesarean Section; Hemodynamic Instability
Keywords: Ceseaean section; Spinal anesthesia; Hemodynamics
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group İzobarik bupivakain (5 mg) + fentanil (Active Comparator): Patients were given a solution containing 5 mg isobaric bupivacaine + 15 µg fentanyl (1.3 ml)
  Interventions: Drug: Bupivacaine
- Group İzobarik bupivakain (7 mg) + fentanil (Active Comparator): Patients were givena solution containing 7 mg isobaric bupivacaine + 15 µg fentanyl (1.7 ml)
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Two Different Low-Doses Of Isobaric Bupivacaine ( Group İzobarik bupivakain (5 mg) + fentanil and Group İzobarik bupivakain (7 mg)+ fentanyl ) were administered to the subarachnoid space

SUMMARY:
The primary aim of this study was to compare the effects of two different low-dose bupivacaine used in spinal anesthesia on intraoperative hemodynamics in cesarean section operations.Investigators think that low-dose bupivacaine and fentanyl mixture applied in cesarean section cause fewer hemodynamic changes,provide adequate anesthesia and analgesia quality,cause fewer side effects,and postoperatively,patients may return to their daily activities more quickly.This study was conducted on 80 pregnant women undergo an elective cesarean section.Patients were randomly allocated in GrupA and GroupB. Combined spinal-epidural anesthesia was performed in the sitting position using the needle-inside-needle technique.After cerebrospinal fluid flow was observed, GroupA patients were given a solution containing 5 mg isobaric bupivacaine+15 µg fentanyl (1.3 ml),and Group B was administered a solution containing 7 mg isobaric bupivacaine+15 µg fentanyl (1.7ml).Hypotension,bradycardia,duration of analgesia,postoperative nausea and vomiting were recorded.

ELIGIBILITY:
Inclusion Criteria

* ASA I-II
* Pregnant women
* 18-50 years of age
* BMI<40kg/m2
* 150-180 cm in height

Exclusion Criteria:

* Patients with hypertension induced by emergency obstetric surgery
* Significant systemic disease,
* Multiple pregnancies,
* Fetal or placental abnormality,
* Hypersensitivity or allergy history to the drugs to be used in the study
* Contraindicated neuraxial anesthesia,
* Infection at or around the region to be anesthetized,
* Coagulation abnormalities
* Patients unable to decide or unwilling to participate in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 80 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
The primary aim of study was to compare the effects of two different low-dose bupivacaine used in spinal anesthesia on intraoperative systolic and diastolic blood pressure (mmHg) in cesarean section operations. | during cesarean procedure
  Intraoperatif hemodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Aksoy, MD, Study Director — Ataturk University, Department of Anesthesiology and Reanimation
Locations (1):
- Aysenur Dostbil, Yakutiye, Erzurum, Turkey (Türkiye)